CLINICAL TRIAL: NCT00861432
Title: Evaluation of Quality of Life of Tumor Patients With and Without Additive Homeopathy.
Brief Title: Evaluation of Questionnaires of Tumor Patients With and Without Additive Homeopathic Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Frass, Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2341
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Tumor
Keywords: Life quality; questionnaire; tumor patients
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- additive homeopathic treatment (Active Comparator): These patients receive additive homeopathic treatment during conventional cancer treatment.
  Interventions: Other: additive homeopathic treatment
- no additive homeopathic treatment (No Intervention): These patients do not receive additive homeopathic treatment during conventional cancer treatment.

INTERVENTIONS:
Other: additive homeopathic treatment — These patients receive additive homeopathic treatment
  Other Names: homeopathic remedies according to the Pharmacopoeia
  Arms: additive homeopathic treatment

SUMMARY:
Tumor patients receiving conventional tumor therapies are included into this study. The patients are randomized into two groups receiving either additive homeopathic therapy or not. Two questionnaires referring to subjective feeling and life quality are filled out by the patients with each visit to the outpatients Department. One of them is the QLQC30 questionnaire of the EORTC. The results of the questionnaires of the two groups are compared.

DETAILED DESCRIPTION:
Quality of life is an important issue for cancer patients, especially during the periods of chemotherapy and radiation. Preliminary results have revealed positive effects of add-on homeopathy on quality of life as well as subjective well-being. Patients are receiving classical homeopathy with administration of either globules and/or dilutions. With each appointment, patients complete two questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Tumor patients between 18 and 100 years old

Exclusion criteria: Patients younger than 18 years, patients having completed less than 3 questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2008-12; Primary Completion 2010-07 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Difference with regard to subjective feeling and life quality with or without homeopathic treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frass, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Med. Univ. Vienna, Dept. Internal Med. I, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frass M, Friehs H, Thallinger C, Sohal NK, Marosi C, Muchitsch I, Gaertner K, Gleiss A, Schuster E, Oberbaum M. Influence of adjunctive classical homeopathy on global health status and subjective wellbeing in cancer patients - A pragmatic randomized controlled trial. Complement Ther Med. 2015 Jun;23(3):309-17. doi: 10.1016/j.ctim.2015.03.004. Epub 2015 Mar 23. PMID 26051564